CLINICAL TRIAL: NCT06114485
Title: Technology-Enabled Services to Support Caregivers of Older Adults With Depression
Brief Title: Voice Activated Personal Assistant for Depression Among Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Allison Carroll, Research Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU#: 00211894
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital Mental Health Intervention (DMHI) (Experimental): Participants randomized to Arm 1 will be sent an Amazon Alexa device, with a newly designed VIPA treatment program installed, and will receive a guidebook to help the older adult understand the device and utilize the VIPA treatment program to its fullest potential.
  Interventions: Behavioral: VIPA Treatment Program
- Control Treatment (CT) (Active Comparator): Participants randomized to Arm 2 will be sent an Amazon Alexa device with guidebook to help the older adult understand how to use the device.
  Interventions: Behavioral: Alexa with Guidebook

INTERVENTIONS:
Behavioral: VIPA Treatment Program — Participants will receive and Alexa device with a behavioral activation program, along with a detailed guidebook about how to utilize the Alexa device and the VIPA program
  Arms: Digital Mental Health Intervention (DMHI)
Behavioral: Alexa with Guidebook — Participants will receive an Alexa device with a detailed guidebook on how to use the device.
  Arms: Control Treatment (CT)

SUMMARY:
Participants will use Amazon Alexa to test a new voice-assisted program for mental health management. The participant will use this program to help with goal setting, reminders, and various other services. The participant may be supported by a caregiver, if available, or by research team member who will serve as a coach for the duration of the study to guide them with using the program. Participants will be asked to complete surveys and assessments about their experiences during the 12-week study period. Participants will be randomized into two groups: those who receive a guide to help them with utilization of the program to its fullest potential and those who do not receive that guide.

DETAILED DESCRIPTION:
Older adults have often been on the fringe of benefiting from technology. However, voice-controlled intelligent personal assistants (VIPAs; e.g. Google Home, Amazon Echo), with their natural interaction style and ease of use, are a simple interface technology that may be useful to older adults with depression in the home setting. The caregiver or coach will be able to schedule and follow the interactions between the older adult and the VIPA. The VIPAs would potentially be able to provide functional, cognitive, and social stimulation as well as improve anti-depressant medication adherence through reminders to older adults.

The aim is to evaluate a VIPA that was designed to deliver behavioral activation prompts to older adults with depression. Through user centered design (UCD), the investigators have adapted the model for remote support with the aid of VIPAs that provide psychoeducation, as well as features that support social, cognitive, and functional stimulation and reminders.

The intervention will be 8 weeks, with a 4-week follow-up. During 8-week intervention, participants will be able to use Amazon Echo Show 8 and the study's VIPA program to set goals, reminders, and the like to help with their mood. Participants will also be asked to completed associated assessments. If caregivers are involved, they will also be asked to complete assessments.

ELIGIBILITY:
Inclusion criteria:

* Adults 65 years or older
* English-speaking
* Elevated depressive symptoms (PHQ-9 ≥ 10)
* Have Wi-Fi access
* Cognitively intact (Montreal Cognitive Assessment (MOCA) score ≥17)

or

Inclusion criteria:

* Adults 18 years or older
* English-speaking
* Provide support to an older adult (65 or older)
* Have access to Wi-Fi
* Demonstrating capacity to consent
* Cognitively intact (Montreal Cognitive Assessment (MOCA) score ≥17 if 65 years or older)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | 12 weeks
  The Patient Health Questionnaire-9 (PHQ-9) PHQ-9 measures depression symptom severity on a scale of 0-27, with higher scores indicating greater symptom severity.
  The PHQ-9 measures depressive symptom severity on a scale of 0-27, with higher scores indicating greater severity
Anxiety symptoms | 12 weeks
  The Generalized Anxiety Disorder-7 (GAD-7) measures anxiety symptom severity on a scale of 0-21, with higher scores indicating greater severity

SECONDARY OUTCOMES:
Adherence | 8 weeks
  The number of times the Alexa device was accessed (Usage; # communications with TES-VIPA)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the NIMH Data Archive
Time Frame: Data will be available 1 year after completion of the study.
Access Criteria: Approval by NIMH Data Archive
URL: https://nda.nih.gov/